CLINICAL TRIAL: NCT00305253
Title: Efficacy Study of the Non-Pneumatic Anti-Shock Garment (NASG) in Egypt
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: MacArthur Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-84956-000-GSS
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hypovolemic Shock; Hemorrhage
Keywords: maternal mortality; obstetric hemorrhage
MeSH Terms: conditions — Shock; Hemorrhage; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-Intervention (No Intervention): The Pre-Intervention Phase served as the Control / Baseline group.
- Post-Intervention (Experimental): Intervention used in this phase and outcomes compared to the Pre-Intervention phase.
  Interventions: Device: Non-pneumatic Anti-shock Garment (NASG)

INTERVENTIONS:
Device: Non-pneumatic Anti-shock Garment (NASG) — In the Post-Intrevention phase of the study, the NASG will be used when a patient meets the study criteria.
  Other Names: NASG; Manufactured by Zoex; Anti-Shock Garment; Life Wrap
  Arms: Post-Intervention

SUMMARY:
This study will test the efficacy of the NASG on women suffering from obstetric hemorrhage as compared to hemorrhaging women who do not receive the NASG.

DETAILED DESCRIPTION:
This is a comparative, pre-post study of the Non-pneumatic Anti-Shock Garment (NASG) to establish its effectiveness in reducing maternal mortality and morbidity due to obstetrical hemorrhage. The sites are two maternity teaching hospitals in Egypt: El Galaa, in Cairo and Assiut University in Assiut.

Our main aim was to test the efficacy of the NASG on women suffering from obstetric hemorrhage as compared to hemorrhaging women who do not receive the NASG. Our primary outcome was Extreme Adverse Outcomes (EAO) - a combined outcome of maternal mortality and severe morbidity. Secondary outcomes included mean measured blood loss and incidence of emergency hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* blood loss from obstetric hemorrhage >= 1000 mL
* pulse > 100 beats per minute or systolic blood pressure < 100 mmHg

Exclusion Criteria:

Absolute exclusion criteria:

* current viable third trimester intrauterine pregnancy that can be delivered in the next 20 minutes after hemorrhage begins
* current bleeding sites above the diaphragm.

Relative exclusion criteria:

* history or current clinical evidence of mitral stenosis or congestive heart failure (CHF)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Miller, CNM, PhD, RN, Principal Investigator — University of California, San Francisco
Locations (2):
- Egypt (2):
  - Assuit University Hospital, Asyut
  - El-Galaa Teaching Hospital, Cairo

REFERENCES:
- [Result] Miller S, Hamza S, Bray EH, Lester F, Nada K, Gibson R, Fathalla M, Mourad M, Fathy A, Turan JM, Dau KQ, Nasshar I, Elshair I, Hensleigh P. First aid for obstetric haemorrhage: the pilot study of the non-pneumatic anti-shock garment in Egypt. BJOG. 2006 Apr;113(4):424-9. doi: 10.1111/j.1471-0528.2006.00873.x. PMID 16553654
- [Result] Miller S, Martin HB, Morris JL. Anti-shock garment in postpartum haemorrhage. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):1057-74. doi: 10.1016/j.bpobgyn.2008.08.008. Epub 2008 Sep 20. PMID 18805742
- [Result] Turan J, Ojengbede O, Fathalla M, Mourad-Youssif M, Morhason-Bello IO, Nsima D, Morris J, Butrick E, Martin H, Camlin C, Miller S. Positive effects of the non-pneumatic anti-shock garment on delays in accessing care for postpartum and postabortion hemorrhage in Egypt and Nigeria. J Womens Health (Larchmt). 2011 Jan;20(1):91-8. doi: 10.1089/jwh.2010.2081. Epub 2010 Dec 29. PMID 21190486
- [Result] Miller S, Fathalla MM, Ojengbede OA, Camlin C, Mourad-Youssif M, Morhason-Bello IO, Galadanci H, Nsima D, Butrick E, Al Hussaini T, Turan J, Meyer C, Martin H, Mohammed AI. Obstetric hemorrhage and shock management: using the low technology Non-pneumatic Anti-Shock Garment in Nigerian and Egyptian tertiary care facilities. BMC Pregnancy Childbirth. 2010 Oct 18;10:64. doi: 10.1186/1471-2393-10-64. PMID 20955600
- [Result] Mourad-Youssif M, Ojengbede OA, Meyer CD, Fathalla M, Morhason-Bello IO, Galadanci H, Camlin C, Nsima D, Al Hussaini T, Butrick E, Miller S. Can the Non-pneumatic Anti-Shock Garment (NASG) reduce adverse maternal outcomes from postpartum hemorrhage? Evidence from Egypt and Nigeria. Reprod Health. 2010 Sep 1;7:24. doi: 10.1186/1742-4755-7-24. PMID 20809942
- [Result] Miller S, Turan JM, Dau K, Fathalla M, Mourad M, Sutherland T, Hamza S, Lester F, Gibson EB, Gipson R, Nada K, Hensleigh P. Use of the non-pneumatic anti-shock garment (NASG) to reduce blood loss and time to recovery from shock for women with obstetric haemorrhage in Egypt. Glob Public Health. 2007;2(2):110-24. doi: 10.1080/17441690601012536. PMID 19280394
- See also: Information and updates on current trials using the Life Wrap (NASG) for obstetric hemorrhage in low resource settings. — http://www.lifewrap.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Intervention: Pre-intervention period: patients experiencing obstetric hemorrhage were treated with standardized evidence-based protocol.
- Post-Intervention: Post-intervention (NASG) period: patients experiencing obstetric hemorrhage were treated with standardized evidence-based protocol plus NASG.
Period: Overall Study
Arm/Group | Pre-Intervention | Post-Intervention
Started | 432 | 559
Completed | 432 | 558
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pre-Intervention: facilities will treat patients with standardized evidence-based protocol when a patient meets the study criteria.
- Post-Intervention: facilities will treat patients with standardized evidence-based protocol plus NASG when a patient meets the study criteria.
- Total: Total of all reporting groups
Arm/Group | Pre-Intervention | Post-Intervention | Total
Number analyzed (Participants) | 432 | 558 | 990
Age Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.2) | 28.9 (6.0) | 28.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 432 | 558 | 990
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 432 | 558 | 990

OUTCOME MEASURES:

1. Primary Outcome: Extreme Adverse Outcomes (EAO) - a Combined Outcome of Maternal Mortality or Severe Morbidity (Cardiac,Respiratory, Renal or Cerebral Dysfunction)
Time Frame: from early pregnancy to within 3 weeks postpartum
Population: All patients enrolled in the study were used in this analysis.
Measure: Number; unit: participants
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 432 | 558
participants | 27 | 11
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Relative risks and confidence intervals were computed for the primary outcome, Extreme Adverse Outcomes (EAO) - a combined measure of maternal mortality or severe mobidity. To estimate the independent effect of the intervention net of the effects of other baseline characteristics, a multiple logistic regression model was used; Test type: Superiority or Other; p = 0.019, Regression, Logistic; Independent variables were selected on the basis of their significant association with EAO in bivariate analyses (t-tests and logistic regression); Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.17 to 0.85] — Pre-Intervention group was compared to the Post-Intervention group. Each group contained different study participants

2. Secondary Outcome: Blood Loss Due to Obstetric Hemorrhage
Description: cumulative blood loss measured hourly upon study admission by calibrated blood collection drape
Time Frame: within 72 hours of study enrollment
Population: Blood loss information was missing on some patients.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 336 | 435
mL | 378.9 (234.3) | 253.2 (205.3)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Mean measured volume of blood loss in the drape was compared across phases with t-tests; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 7.79 — Pre-Intervention group was compared to the Post-Intervention group. Each group contained different study participants

3. Secondary Outcome: Emergency Hysterectomy
Description: incidence of emergency hysterectomy for cases of uterine atony
Time Frame: within 72 hours of study enrollment
Population: Data on emergency hysterectomy are only for women with diagnosis of uterine atony.
Measure: Number; unit: participants
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 278 | 396
participants | 35 | 28
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Relative risks and confidence intervals were computed for emergency hysterectomy; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Risk Ratio (RR) = 0.41, 95% CI 2-sided [0.21 to 0.80] — Pre-Intervention group was compared to the Post-Intervention group. Each group contained different study participants

ADVERSE EVENTS:
Arm/Group | Pre-Intervention | Post-Intervention
Serious Adverse Events (participants affected / at risk) | 10/432 | 6/558
Other Adverse Events (participants affected / at risk) | 17/432 | 5/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Intervention (N=432) | Post-Intervention (N=558)
Mortality (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Intervention (N=432) | Post-Intervention (N=558)
Renal Failure (Renal and urinary disorders) | 14 (14) | 3 (3) — Other adverse events are all designated as morbidities in publications. Three individuals in the pre-intervention group suffered two other adverse events each, but in analysis are considered single morbidities.
Acute Respitory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cerebral Impairment (Nervous system disorders) | 2 (2) | 2 (2)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Non-randomized, non-blinded pre-intervention/intervention design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Local PIs are required to review results with Dr. Miller before releasing.